CLINICAL TRIAL: NCT05376839
Title: A Phase 1 Study to Evaluate the Pharmacokinetics and Safety of Multiple Doses of Cedirogant (ABBV-157) in Subjects With Mild, Moderate and Severe Hepatic Impairment
Brief Title: A Study to Assess Safety of Cedirogant and How Cedirogant Moves Through the Body in Adult Participants With Mild, Moderate and Severe Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-367
Record Dates: First submitted 2022-05-13; First posted 2022-05-17 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hepatic Impairment
Keywords: Cedirogant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Cedirogant (Experimental): Participants will receive cedirogant once daily.
  Interventions: Drug: Cedirogant
- Group 2: Cedirogant (Experimental): Participants will receive cedirogant once daily.
  Interventions: Drug: Cedirogant
- Group 3: Cedirogant (Experimental): Participants will receive cedirogant once daily.
  Interventions: Drug: Cedirogant
- Group 4: Cedirogant (Experimental): Participants will receive cedirogant once daily.
  Interventions: Drug: Cedirogant

INTERVENTIONS:
Drug: Cedirogant — Capsule, Oral

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics and safety of cedirogant following oral administration of multiple doses in adult participants with hepatic impairment and normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is ≥ 18.0 to < 40 kg/m2
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile (except liver function tests for subjects with hepatic impairment), and 12-lead ECG

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests (except liver function tests for subjects with hepatic impairment) at screening that is assessed as likely to interfere with the objectives of the trial or the safety of the subject.
* History or evidence of active TB or latent TB infection
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of cervix

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 18 Days
  Maximum Observed Plasma Concentration
Time to maximum observed plasma concentration (Tmax) | Up to 18 Days
  Time to maximum observed plasma concentration
Area under the plasma concentration-time curve (AUC) from time 0 to 24 hours after dosing (AUC0-24) | Up to 18 Days
  AUC from time 0 to 24 hours after dosing

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Up to 44 Days
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami /ID# 246573, Miami, Florida
  - Orlando Clinical Research Ctr /ID# 246052, Orlando, Florida
  - TX Liver Inst, Americ Res Corp /ID# 246572, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No